CLINICAL TRIAL: NCT01802489
Title: A Double Blind Randomised Control Trial on Neuroprotection of Amiloride in Optic Neuritis
Brief Title: Amiloride Clinical Trial In Optic Neuritis
Acronym: ACTION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Multiple Sclerosis Society of Great Britain and Northern Ireland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Amiloride 02
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Optic Neuritis; Multiple Sclerosis
Keywords: Optic neuritis; Multiple sclerosis; Retinal nerve fibre layer; Axonal loss; Neuroprotection; MRI; Optical coherence tomography; Amiloride; Acid Sensing Ion Channels
MeSH Terms: conditions — Optic Neuritis; Multiple Sclerosis | interventions — Amiloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amiloride (Active Comparator): Amiloride capsules 10mg once per day for 5 months
  Interventions: Drug: Amiloride
- Placebo (Placebo Comparator): Placebo capsules one per day for 5 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amiloride
  Other Names: Midamor
  Arms: Amiloride
Drug: Placebo — Placebo capsule identical in appearance to Amiloride 10mg capsule
  Arms: Placebo

SUMMARY:
Optic neuritis (ON) is a common event in Multiple Sclerosis (MS), and causes significant loss of nerve cells in the eye, resulting in poor vision. Optic neuritis also provides a sensitive way of testing the effectiveness of drugs that may help protect from loss of nerve cells in ON and therefore in MS.

The investigators have identified through laboratory and early clinical research in humans that amiloride (a water tablet already in use) may be a drug that can be of benefit in optic neuritis by protecting from loss of nerves cells, ie a neuroprotective drug.

The purpose of this study is to assess the efficacy of amiloride as a neuroprotective drug in optic neuritis

DETAILED DESCRIPTION:
Multiple sclerosis (MS), an inflammatory condition of the nervous system, is the most common cause of disability in people of working age in the western world. In addition to the inflammatory episodes in MS, axonal and neuronal damage occurs. It is this axonal loss which is thought to be the major pathological substrate for disability in MS.

Acute inflammatory demyelinating optic neuritis is a common event in multiple sclerosis. Following optic neuritis there is axonal loss in the optic nerve and retina, which if severe can result in a poor visual recovery. Uniquely amongst central nervous system (CNS) structures, the structural and functional changes in the eye during and following optic neuritis provide a sensitive way of observing neurodegeneration and testing the effectiveness of potential neuroprotective agents. In optic neuritis it has been shown that thinning of the retinal nerve fibre layer takes place, and by 6 months this thinning is established and has largely stabilised. This represents axonal loss in the anterior visual system. The degree of this thinning has been shown to correlate with the amount of vision recovered following optic neuritis, the more thinning that occurs, the poorer the outcome. The thickness of the retinal nerve fibre layer can be measured by the simple scanning techniques of scanning laser polarimetry (GDx) and optical coherence tomography (OCT).

Axonal loss in MS is likely to be multifactorial, but a key end point is the influx of sodium and calcium ions. Recent research suggests that in the inflammatory environment of optic neuritis, the acid sensing ion channel may have an important role in this influx of sodium and calcium, and therefore in axonal loss in MS. The drug amiloride, already in use as a diuretic, is a known blocker of this ion channel. The investigators have identified through laboratory and early clinical research in humans that by blockade of the acid sensing ion channel, amiloride may be neuroprotective in optic neuritis and MS.

The investigators primary objective is to assess the neuroprotective efficacy of amiloride in optic neuritis through the surrogate measure of retinal nerve fibre layer measurement. Secondary objectives are to assess markers of neurodegeneration in ON and the neuroprotective effect of amiloride through non-conventional MRI outcomes, to assess if amiloride improves functional and visual outcome following optic neuritis, and to confirm optic neuritis as a sensitive and efficient model for neuroprotection in a clinical trial framework.

46 Participants will be recruited to receive either amiloride, or an identical placebo capsule for 5 months. The primary outcome will be measured at 6 months, with a further measure at 12 months.

Should this trial show a significant benefit from amiloride in optic neuritis, it will be an important first step in developing neuroprotective therapies in optic neuritis and MS and potentially this could have a significant impact on people with MS and their carers.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a first episode of unilateral optic neuritis
* Participants with an existing diagnosis of relapsing remitting MS and new onset of ON are eligible if they have;

  1. Not had a previous episode of optic neuritis,
  2. A duration of disease of ≤10 years
  3. An EDSS (Expanded Disability Status Scale) of ≤3.
  4. No immune modulating treatment other than β-Interferon or glatiramer acetate at time of recruitment
* Able to be randomised within 28 days of onset of visual symptoms
* Visual acuity of ≤6/9
* Participant is willing and able to give informed consent for participation in the study and able to comply with study visits
* Male or Female, aged between18 - 55 years.
* Stable dose of current regular medication for at least 4 weeks prior to study entry.
* Participant has clinically acceptable urea and electrolytes and estimated glomerular filtration rate (eGFR) >60
* Able and willing to comply with all study requirements.
* Willing to allow his or her General Practitioner to be notified of participation in the study.

Exclusion Criteria:

* Previous diagnosis of optic neuritis
* Any concomitant immune suppressing or immune modulating therapy excluding β-interferon or glatiramer acetate.
* Female participants who are pregnant, lactating or planning pregnancy during the course of the study.
* Concomitant potassium supplements, angiotensin converting enzyme inhibitors, angiotensin II antagonists, cyclosporine, tacrolimus or lithium
* Any contra-indication to MRI - severe claustrophobia, metal implant, pacemaker, etc.
* Participant who is terminally ill or is inappropriate for placebo medication
* Impaired renal function : eGFR ≤60, anuria, acute or chronic renal insufficiency and evidence of diabetic nephropathy
* Raised serum potassium (K+ >5.5mmol/l)
* Diabetes
* Significant concomitant eye disease in either eye that may affect diseased or fellow eye results.
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Participants who have participated in another research study involving an investigational product in the past 12 weeks.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2013-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Scanning laser polarimetry determined retinal nerve fibre layer thickness | Baseline, 6 and 12 months
  The primary outcome will be difference in retinal nerve fibre thickness at 6 months between affected eye and non-affected fellow eye at baseline between the amiloride and placebo group.
  An additional measure will be made at 12 months

SECONDARY OUTCOMES:
Optical coherence tomography determined difference in retinal nerve fibre layer thickness. | Baseline, 6 and 12 months
  Difference in thickness at 6 months and 12 months between affected eye and non-affected fellow eye at baseline, between the amiloride and placebo group
Differences between the amiloride and placebo groups in non-conventional MRI surrogate marker of white matter and grey matter injury and connectivity by 3T scanning. | Baseline, 6 and 12 months
  * Diffusion weighted imaging (DWI) - measures; fractional anisotropy (FA), mean diffusivity (MD), axial and radial diffusivity (RD) of the posterior visual tracts
  * High Resolution T1-weighted image measure of grey matter volume
  * Magnetic resonance spectroscopy (MRS) measures of N-acetyl aspartate (NAA) in the visual cortex
  * Resting state functional MRI (RS fMRI) patterns of activity
  * Magnetisation transfer imaging (MTI) derived magnetisation transfer ratio (MTR) of the white and grey matter
Visual Function | Baseline, 6 and 12 months
  * High and low contrast (2.5% and 1.25%) visual acuity.
  * Farnsworth Munsell 100 Hue (FM100) colour vision test.
Visual Electrophysiology | 0 and 6 months
  Differences in visually evoked potential and pattern electro-retinogram between the amiloride and placebo groups as additional measures of visual function
Quality of life questionnaires | Baseline, 6 and 12 months
  * 25 point national institutes for health visual function questionnaire
  * 10 point neuro ophthalmic supplement.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Craner, MBChB PhD, Principal Investigator — University of Oxford
Locations (1):
- John Radcliffe Hospital, Oxford, United Kingdom

REFERENCES:
- [Derived] McKee JB, Cottriall CL, Elston J, Epps S, Evangelou N, Gerry S, Kennard C, Kong Y, Koelewyn A, Kueker W, Leite MI, Palace J, Craner M. Amiloride does not protect retinal nerve fibre layer thickness in optic neuritis in a phase 2 randomised controlled trial. Mult Scler. 2019 Feb;25(2):246-255. doi: 10.1177/1352458517742979. Epub 2017 Nov 27. PMID 29172994
- [Derived] McKee JB, Elston J, Evangelou N, Gerry S, Fugger L, Kennard C, Kong Y, Palace J, Craner M. Amiloride Clinical Trial In Optic Neuritis (ACTION) protocol: a randomised, double blind, placebo controlled trial. BMJ Open. 2015 Nov 9;5(11):e009200. doi: 10.1136/bmjopen-2015-009200. PMID 26553836